CLINICAL TRIAL: NCT04899505
Title: ODORAJA:Evaluation of the Impact of Chemotherapy on Body Odor in Adolescents and Young Adults in Oncology
Brief Title: Evaluation of the Impact of Chemotherapy on Body Odor in Adolescents and Young Adults in Oncology
Acronym: ODORAJA
Status: Completed | Type: Observational
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Other Study IDs: IC 2021-02
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2023-01

CONDITIONS: Solid Tumor, Adult; Solid Tumor, Childhood; Chemotherapy Effect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Evaluation on appearance of unpleasant body odors: Incidence of the development of unpleasant body odors in AYA oncology patients
  Interventions: Other: Evaluation on appearance of unpleasant body odors

INTERVENTIONS:
Other: Evaluation on appearance of unpleasant body odors — Percentage of patients reporting discomfort with unpleasant body odor that occurred during their treatment. This percentage will be calculated from the response to item Q1 of the patient questionnaire during the fourth course of chemotherapy in the AJA oncology department.

SUMMARY:
The appearance of unpleasant body odors in adolescent Young adult (aya) wille be evaluated undergoing chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 15 and 25 years;
* New patients treated at the Curie Institute and hospitalized in the AJA oncology department;
* Patient undergoing chemotherapy administered intravenously;
* Solid tumors.

Exclusion Criteria:

* Patient undergoing oral chemotherapy;
* Persons deprived of their liberty or under guardianship (including guardianship);
* Inability to undergo medical monitoring of the trial for geographical, social or psychological reasons.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients aged between 15 and 25 years with solid tumors
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Incidence of the development of unpleasant body odors in AYA oncology patients | 8 months
  Percentage of patients reporting discomfort with unpleasant body odor that occurred during their treatment. This percentage will be calculated from the response to item Q1 of the patient questionnaire during the fourth course of chemotherapy in the AJA oncology department

SECONDARY OUTCOMES:
Qualification of the smell and the discomfort felt | 8 months
  Answers to the investigation intended for patients for the appearance of the smell with different proposals like sweating, urine, breath etc. (Q2), its qualifier with different proposals like desagreable, infective, nauseating, etc…(Q3) and the discomfort observed for themselves or for those around them (Q8)
Quantification of the discomfort and the impact on quality of life | 8 months
  Answers to the investigation intended for patients to assess the intensity of the smell with a scale (0= no smell and 10 = strong smell) (Q4), its daily impact with a scale (0=no impact and 10= high impact) (Q7) and solutions that can reduce smell with different proposals like perfume, cream, essential oil (Q9)
Identify possible causes of the appearance of these new body odors | 8 months
  Answers to the investigation for patients to assess the link between smell and drug treatment with different proposals like treatment, hospital's food or hospital cleaning product (Q5 and Q6)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Curie, Paris, France